CLINICAL TRIAL: NCT00005941
Title: Phase II Pilot Trial of Non-Myeloablative Allogeneic Peripheral Blood Stem Cell (PBSC) Transplantation Using Fludarabine, Low Dose TBI and Post-Transplant Cyclosporine and Mycophenolate Mofetil Followed by Donor Lymphocyte Infusion for Therapy of Advanced or Metastatic Human Papilloma Virus (HPV) - Associated Cervical Carcinoma Refractory to Standard Therapy
Brief Title: Peripheral Stem Cell Transplant, White Blood Cell Infusions, Chemotherapy, and Radiation Therapy in Treating Patients With Recurrent Metastatic Cervical or Vaginal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1477.00; FHCRC-1477.00; NCI-G00-1784; CDR0000067816 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-03

CONDITIONS: Cervical Cancer; Vaginal Cancer
Keywords: stage III cervical cancer; recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vaginal cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — Cyclosporine; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: mycophenolate mofetil
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving low doses of chemotherapy, such as fludarabine, and radiation therapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well donor peripheral stem cell transplant plus chemotherapy and total-body irradiation followed by donor white blood cell infusion work in treating patients with recurrent metastatic or locally advanced cancer of the cervix or vagina that is associated with human papillomavirus.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the partial or complete response in patients with recurrent metastatic or locally advanced human papillomavirus (HPV)-associated cervical or vaginal carcinoma treated with a nonmyeloablative regimen comprising fludarabine and low-dose total body irradiation followed by allogeneic peripheral blood stem cell transplantation, cyclosporine, mycophenolate mofetil, and donor lymphocyte infusion.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine whether this regimen induces engraftment and donor chimerism in these patients.
* Determine the HPV-E6 and HPV-E7 specific T-cell responses in selected patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients receive conditioning therapy comprising fludarabine IV on days -4 to -2 and low-dose total body irradiation on day 0. Filgrastim (G-CSF)-mobilized allogeneic peripheral blood stem cells are infused on day 0.

Patients also receive oral cyclosporine twice daily on days -3 to 35 and then tapered until day 56. Mycophenolate mofetil is administered orally twice daily on days 0-27.

Patients with disease progression and no graft-versus-host disease on day 56 receive nonmobilized donor lymphocyte infusion (DLI) over 30 minutes on day 65. DLI may be repeated every 65 days for up to 4 doses.

Patients are followed weekly for 3 months, monthly for 6 months, every 6 months for 2 years, and then annually for 5 years.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent metastatic or locally advanced cervical or vaginal carcinoma that is not curable with surgery or radiotherapy

  * Tumor is human papillomavirus positive by polymerase chain reaction
* Bidimensionally measurable disease by clinical examination or radiographic imaging
* Availability of an genotypically HLA-identical sibling donor (excluding identical twins)
* No brain metastases

PATIENT CHARACTERISTICS:

Age:

* Under 65

Performance status:

* Karnofsky 80-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN

Renal:

* Creatinine clearance at least 40 mL/min

Cardiovascular:

* Cardiac ejection fraction at least 40%
* No history of congestive heart failure
* No poorly controlled hypertension

Pulmonary:

* No severe defects in pulmonary function
* No supplementary continuous oxygen

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 12 months after study completion
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Concurrent growth factors for severe persistent or febrile neutropenia after transplantation allowed

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Max Age: 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1999-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Partial or complete response

SECONDARY OUTCOMES:
Toxicity
Engraftment and donor chimerism
HPV-E6 and E7-specific T cell responses

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nash, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States